CLINICAL TRIAL: NCT04865536
Title: A Phase 1, Partially-Blinded, Placebo-Controlled, Randomized, Multiple Ascending Dose Study to Include A Single Dose Food-Effect Study to Evaluate the Safety, Tolerability, and the PK Profile of TBI-223 in Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability, and the PK Profile of TBI-223 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TBI-223-CL-002
Record Dates: First submitted 2021-02-22; First posted 2021-04-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
Keywords: TB; Tuberculosis; TBI-223; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TBI-223 1800 mg (Active Comparator): Cohort 1, 3 x 600 mg slow release (SR1) tablets. Administered on Day 1 under fasted conditions, followed by a 3-day washout period and then by multiple doses of TBI-223 administered after a high-calorie, high-fat meal (Fed) from Day 4 through Day 17 (total of 14 days), (n=9)
  Interventions: Drug: TBI-223 1800 mg
- TBI-223 2400mg (Active Comparator): Cohort 2, 3 x 600 mg SR1 tablets and 1 x 600 mg immediate release (IR) tablets. Administered on Day 1 under fasted conditions, followed by a 3-day washout period and then by multiple doses of TBI-223 administered after a high-calorie, high-fat meal (Fed) from Day 4 through Day 17 (total of 14 days), (n=13)
  Interventions: Drug: TBI-223 2400mg
- TBI-223 Placebo (Placebo Comparator): Dose matching placebo tablets. Administered on Day 1 under fasted conditions, followed by a 3-day washout period and then by multiple doses of dose matched placebo administered after a high-calorie, high-fat meal (Fed) from Day 4 through Day 17 (total of 14 days), (n=6)
  Interventions: Drug: TBI-223 Placebo

INTERVENTIONS:
Drug: TBI-223 1800 mg — 3 x 600 mg SR1 tablets
  Arms: TBI-223 1800 mg
Drug: TBI-223 2400mg — 3 x 600 mg SR1 tablets and 1 x 600 mg IR tablets
  Arms: TBI-223 2400mg
Drug: TBI-223 Placebo — Placebo SR and IR tablets for TBI-223
  Arms: TBI-223 Placebo

SUMMARY:
A Phase 1, Partially-Blinded, Placebo-Controlled, Randomized, Multiple Ascending Dose Study to Include A Single Dose Food-Effect Study to Evaluate the Safety, Tolerability, and the PK Profile of TBI-223 in Healthy Subjects

DETAILED DESCRIPTION:
This study was a partially-blinded, placebo-controlled, randomized multiple ascending dose (MAD) study conducted at one study center. Cohorts 1 (1800 mg) and 2 (2400mg) began dosing of TBI-223 or placebo on Day 1 under fasted conditions, followed by a 3-day washout period and then by multiple doses of TBI-223 administered after a high-calorie, high-fat meal (Fed) from Day 4 through Day 17 (total of 14 days). Cohort 1 subjects only received slow-release formulations (SR1) tablets and Cohort 2 subjects received a combination of SR1 tablets with one immediate-release (IR) tablet. Cohort 3 with higher doses was planned in the protocol but as allowed by the protocol, a decision was made to halt the study after the second cohort due to mean Cmax and AUC0-24 after 14 days of dosing at 2400 mg in the second cohort exceeded values that were predicted to be achieved at 3000 mg in the third cohort.

Safety was assessed throughout the study for all subjects. Safety assessments included physical and detailed neurological examinations, vital signs (blood pressure (BP), pulse rate (PR), respiration rate, temperature, and pulse oximetry), 12-lead electrocardiograms (12-lead ECGs), cardiac monitoring, adverse events (AEs), and clinical laboratory tests (including hematology, serology, serum chemistry, coagulation, and urinalysis).

ELIGIBILITY:
Key Inclusion Criteria:

All volunteers must satisfy the following criteria to be considered for study participation:

1. Is a healthy adult male or female, 19 to 50 years of age (inclusive) at the time of screening.
2. Has a body mass index (BMI) ≥18.5 and ≤32.0 (kg/m2) and a body weight of no less than 50.0 kg.
3. Is medically healthy with no clinically significant screening results (e.g., laboratory profiles normal or up to Grade 1 per Division of Microbiology and Infectious Diseases Toxicity Tables), as deemed by the Investigator.
4. Has not used tobacco- or nicotine-containing products (including smoking cessation products), for a minimum of 6 months before dosing.
5. If assigned to receive study drug under fed conditions, is willing and able to consume the entire high-calorie, high-fat breakfast meal in the timeframe required.

Key Exclusion Criteria:

1. History or presence of clinically significant cardiovascular (heart murmur), pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
2. Any presence of musculoskeletal toxicity (severe tenderness with marked impairment of activity, or frank necrosis).
3. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV at screening.
4. QTcF interval >450 msec for males or >470 msec for females at screening, Day -1, or Day 1 (predose), or history of prolonged QT syndrome. For the triplicate 12-lead ECGs taken at screening and on Day -1, the average QTcF interval of the three 12-lead ECG recordings were used to determine qualification.
5. Family history of long-QT syndrome or sudden death without a preceding diagnosis of a condition that was causative of sudden death (such as known coronary artery disease, congestive heart failure, or terminal cancer).
6. History of any of the following:

   * Serotonin syndrome
   * Seizures or seizure disorders, other than childhood febrile seizures
   * Brain surgery
   * History of head injury in the last 5 years
   * Any serious disorder of the nervous system particularly one that lowered the seizure threshold.
7. Lactose intolerant.
8. History of sensitivity or contraindication to use of linezolid, tedizolid, or any study investigational products

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Safety assessment Vital Signs - Blood pressure | through study completion, 12 weeks.
  Blood pressure measured.
Safety assessment Vital Signs - Pulse rate | through study completion, 12 weeks.
  Pulse rate measured.
Safety assessment Vital Signs - Respiration rate | through study completion, 12 weeks.
  Respiration rate measured.
Safety assessment Vital Signs - Temperature | through study completion, 12 weeks.
  Temperature measured.
Safety assessment Vital Signs - Pulse oximetry | through study completion, 12 weeks.
  Pulse oximetry measured.
Safety assessment - Cardiac monitoring | through study completion, 12 weeks.
  Safety 12-lead ECGs including ECG QT interval will be recorded and printed for on-site review by the Principal Investigator or designee.
Safety assessment - Adverse Events (AEs) | through study completion, 12 weeks.
  AEs recorded.
Safety assessment Clinical Laboratory Tests - Hematology | through study completion, 12 weeks.
  Hematology recorded: hemoglobin, hematocrit, total and differential leukocyte count, red blood cell count (RBC), and platelet count.
Safety assessment Clinical Laboratory Tests - Serology | through study completion, 12 weeks.
  Serology tests recorded: hepatitis B surface antigen, hepatitis C antibody, and HIV.
Safety assessment Clinical Laboratory Tests - Serum Chemistry | through study completion, 12 weeks.
  Serum chemistry recorded: albumin, blood urea nitrogen (BUN), creatinine, total bilirubin, alkaline phosphatase (ALP), aspartate transaminase (AST), alanine transaminase (ALT), sodium (Na+), potassium (K+), chloride (Cl-), lactate dehydrogenase (LDH), calcium (Ca), uric acid, glucose, gamma-glutamyltransferase (GGT), and magnesium.
Safety assessment Clinical Laboratory Tests - Coagulation | through study completion, 12 weeks.
  Coagulation recorded: prothrombin time (PT), partial thromboplastin time (PTT), and international normalized ratio (INR).
Safety assessment Clinical Laboratory Tests - Urinalysis | through study completion, 12 weeks.
  Urinalysis recorded.
Safety assessment - Serum Pregnancy Testing | through study completion, 12 weeks.
  Blood collection from female subjects for serum pregnancy testing.
Safety assessment - Follicle-stimulating hormone (FSH) Levels | through study completion, 12 weeks.
  Blood collection from postmenopausal women to measure FSH levels.
Pharmacokinetics, non-food-effect cohorts - AUCtau | Day 1
  AUCtau measured.
Pharmacokinetics, non-food-effect cohorts - Cmax | Day 1
  Cmax measured.
Pharmacokinetics, non-food-effect cohorts - C24 | Day 1
  C24 measured.
Pharmacokinetics, non-food-effect cohorts - Cavg | Day 1
  Cavg measured.
Pharmacokinetics, non-food-effect cohorts - Tmax | Day 1
  Tmax measured.
Pharmacokinetics, non-food-effect cohorts - AUCinf | Day 1
  AUCinf measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, non-food-effect cohorts - AUCextrap | Day 1
  AUCextrap measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, non-food-effect cohorts - CL/F | Day 1
  CL/F measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, non-food-effect cohorts - Vz/F | Day 1
  Vz/F measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, non-food-effect cohorts - lambaZ | Day 1
  lambaZ measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, non-food-effect cohorts - t1/2 | Day 1
  t1/2 measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, non-food-effect cohorts - AUCtau | Day 14
  AUCtau measured.
Pharmacokinetics, non-food-effect cohorts - Cmax | Day 14
  Cmax measured.
Pharmacokinetics, non-food-effect cohorts - Cmin | Day 14
  Cmin measured.
Pharmacokinetics, non-food-effect cohorts - Ctrough | Day 14
  Ctrough (i.e., C0) measured.
Pharmacokinetics, non-food-effect cohorts - C24 | Day 14
  C24 measured.
Pharmacokinetics, non-food-effect cohorts - Cavg | Day 14
  Cavg measured.
Pharmacokinetics, non-food-effect cohorts - Tmax | Day 14
  Tmax measured.
Pharmacokinetics, non-food-effect cohorts - CL/F | Day 14
  CL/F measured.
Pharmacokinetics, non-food-effect cohorts - Vz/F | Day 14
  Vz/F measured.
Pharmacokinetics, non-food-effect cohorts - lambaZ | Day 14
  lambaZ measured.
Pharmacokinetics, non-food-effect cohorts - t1/2 | Day 14
  t1/2 measured.
Pharmacokinetics, non-food-effect cohorts - RAUC | Day 14
  RAUC measured.
Pharmacokinetics, non-food-effect cohorts - RCmax measured. | Day 14
  RCmax measured.
Pharmacokinetics, food-effect cohorts - AUCtau | Day 1
  AUCtau measured.
Pharmacokinetics, food-effect cohorts - AUCextrap | Day 1
  AUCextrap measured.
Pharmacokinetics, food-effect cohorts - AUCinf | Day 1
  AUCinf measured.
Pharmacokinetics, food-effect cohorts - Cmax | Day 1
  Cmax measured.
Pharmacokinetics, food-effect cohorts - C24 | Day 1
  C24 measured
Pharmacokinetics, food-effect cohorts - Clast | Day 1
  Clast measured.
Pharmacokinetics, food-effect cohorts - Tmax | Day 1
  Tmax measured.
Pharmacokinetics, food-effect cohorts - Tlast | Day 1
  Tlast measured.
Pharmacokinetics, food-effect cohorts - CL/F | Day 1
  CL/F measured.
Pharmacokinetics, food-effect cohorts - Vz/F | Day 1
  Vz/F measured.
Pharmacokinetics, food-effect cohorts - lambaZ | Day 1
  lambaZ measured.
Pharmacokinetics, food-effect cohorts - t1/2 | Day 1
  t1/2 measured.
Pharmacokinetics, food-effect cohorts - AUCtau | Day 4
  AUCtau measured. lambaZ, t1/2 should be included if AUCtau ≥ 70% of AUCinf
Pharmacokinetics, food-effect cohorts - Cmax | Day 4
  Cmax measured.
Pharmacokinetics, food-effect cohorts - C24 | Day 4
  C24 measured.
Pharmacokinetics, food-effect cohorts - Cavg | Day 4
  Cavg measured.
Pharmacokinetics, food-effect cohorts - Tmax | Day 4
  Tmax measured.
Pharmacokinetics, food-effect cohorts - AUCinf | Day 4
  AUCinf measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, food-effect cohorts - AUCextrap | Day 4
  AUCextrap measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, food-effect cohorts - CL/F | Day 4
  CL/F measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, food-effect cohorts - Vz/F | Day 4
  Vz/F measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, food-effect cohorts - lambaZ | Day 4
  lambaZ measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, food-effect cohorts - t1/2 | Day 4
  t1/2 measured if AUCtau ≥ 70% of AUCinf.
Pharmacokinetics, food-effect cohorts - AUCtau | Day 17
  AUCtau measured.
Pharmacokinetics, food-effect cohorts - Cmax | Day 17
  Cmax measured.
Pharmacokinetics, food-effect cohorts - Cmin | Day 17
  Cmin measured.
Pharmacokinetics, food-effect cohorts - Ctrough | Day 17
  Ctrough (i.e., C0) measured.
Pharmacokinetics, food-effect cohorts - C24 | Day 17
  C24 measured.
Pharmacokinetics, food-effect cohorts - Cavg | Day 17
  Cavg measured.
Pharmacokinetics, food-effect cohorts - Tmax | Day 17
  Tmax measured.
Pharmacokinetics, food-effect cohorts - CL/F | Day 17
  CL/F measured.
Pharmacokinetics, food-effect cohorts - Vz/F | Day 17
  Vz/F measured.
Pharmacokinetics, food-effect cohorts - lambaZ | Day 17
  lambaZ measured.
Pharmacokinetics, food-effect cohorts - t1/2 | Day 17
  t1/2 measured.
Pharmacokinetics, food-effect cohorts - RAUC | Day 17
  RAUC measured.
Pharmacokinetics, food-effect cohorts - RCmax | Day 17
  RCmax measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Nedelman, Study Chair — Global Alliance for TB Drug Development
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

REFERENCES:
- [Result] Lombardi A, Pappas F, Bruinenberg P, Nedelman J, Taneja R, Hickman D, Beumont M, Sun E. Pharmacokinetics, tolerability, and safety of TBI-223, a novel oxazolidinone, in healthy participants. Antimicrob Agents Chemother. 2025 Apr 2;69(4):e0154224. doi: 10.1128/aac.01542-24. Epub 2025 Mar 11. PMID 40067046

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT04865536/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT04865536/SAP_001.pdf